CLINICAL TRIAL: NCT05804812
Title: The Effect of Laughter Therapy in Women With Migraine
Brief Title: The Effect of Laughter Therapy in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sinop University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: sinopUmeryem-2
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-03

CONDITIONS: Migraine; Laughter
Keywords: migraine; laughter therapy; young women
MeSH Terms: conditions — Migraine Disorders; Laughter | interventions — Laughter Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): At the beginning of the study, data collection tools Personal Information Form and Psychological Well-Being Scale will be applied to the control group.
  No intervention will be made in the control group. Measurement tools will be applied for the post-test.
- experimental group (Experimental): Inclusion criteria for the research: Faculty of Health Sciences, to study in the 2022-2023 academic spring semester, to have been diagnosed with migraine, to be young and to volunteer to participate in the research. Exclusion criteria from the study; Not studying at the Faculty of Health Sciences and not volunteering to participate in the research. The application and control group will be determined on random.org among the group that constitutes the sample of the study. Laughter therapy sessions will be applied online for 25-30 minutes once a week for 2 months by the researcher who has the Laughter therapy certificate to the application group. At the end of two months, the Personal Information Form and Psychological Well-Being Scale will be administered again to both the application group and the control group.
  Interventions: Behavioral: laughter therapy

INTERVENTIONS:
Behavioral: laughter therapy — Assigned Interventions Laughter therapy session will be applied online for 25-30 minutes once a week for 2 months by the researcher who has the Laughter therapy certificate to the application group. In the laughter therapy session, the practices of introducing the practitioner and introducing the therapy, breathing exercises for a healthy life, keeping the rhythm accompanied by music, turning the laughter that started as if it were childlike games into reality will be carried out.
  Arms: experimental group

SUMMARY:
Migraine: An episodic disorder consisting of severe headache, usually with photophobia (sensitivity to light), phonophobia (sensitivity to sound), and/or nausea (occasionally vomiting). Migraine is predominantly a female disease. The incidence of migraine was found to in women (18.2/1000 person-years) and between the ages of 15-19 in men (6.2/1000 person-years). The incidence of migraine was found to peak between the ages of 20-24 in women (18.2/1000 person-years) and between the ages of 15-19 in men (6.2/1000 person-years). Migraine treatments are generally classified as pharmacological (treatment with medication) and non-pharmacological (treatment with no medication). Laughter therapy has recently come to the fore as a non-pharmacological and alternative treatment in chronic pain management. In a randomized controlled study, 30 minutes of laughter therapy was applied to women on the 2nd and 6th days after mastectomy surgery and it was determined that women who received laughter therapy had a significant decrease in pain and anxiety levels. This study was planned to determine the effect of laughter therapy on women with migraine.

DETAILED DESCRIPTION:
The research will be carried out with young girls who are studying at the Faculty of Health Sciences of Sinop University in the 2022-2023 academic spring semester. Inclusion criteria for the research: Faculty of Health Sciences, to study in the 2022-2023 academic spring semester, to have been diagnosed with migraine, to be young girls and to volunteer to participate in the research. Exclusion criteria from the study; Not studying at the Faculty of Health Sciences and not volunteering to participate in the research. The application and control group will be determined on random.org among the group that constitutes the sample of the study. Laughter therapy sessions will be applied online for 25-30 minutes once a week for 2 months by the researcher who has the Laughter therapy certificate to the application group. At the end of two months, the Personal Information Form and Psychological Well-Being Scale will be administered again to both the application group and the control group.

ELIGIBILITY:
Inclusion Criteria:

* Being a nursing student,
* Being a female student,
* Volunteering to participate in the study.
* Being a woman
* Being diagnosed with migraine

Exclusion Criteria:

* Not to study as a nursing student

  * Being a male student
  * Not to volunteer to participate in the study
  * Not being a woman between the ages of 18 and 30

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 53 (Actual)
Dates: Start 2023-04-06 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
1. Personal İnformation form | one day
  Personal İnformation form consists of 2 parts. In the first part, the socio-demographic characteristics of the individual, such as class, age, place and region where he lives the longest, mother and father working status, economic status, consist of 9 questions. In the second part, it consists of a total of 9 questions about the characteristics of migraine, including migraine location, frequency, duration of attendance, duration of medication, severity, coping methods, complaints associated with migraine, time without medication, and school attendance.

SECONDARY OUTCOMES:
2. Psychological Well-Being Scale: | one day
  The Psychological Well-Being Scale was developed by Diener et al. (2009-2010) to measure socio-psychological well-being, complementary to existing well-being measures. The Turkish adaptation of the scale was done by Telef (2011; 2013). It was determined that the item-total correlations of the Psychological Well-Being Scale varied between .41 and .63, and the t-values were significant (p<.001). The items of the Psychological Well-Being Scale are answered between 1 and 7, as I strongly disagree (1) to I strongly agree (7). All items are expressed positively. Scores range from 8 (strongly disagree to all items) to 56 (strongly agree to all items).

CONTACTS AND LOCATIONS:
Overall Officials: Meryem Erdoğan, PhD, Principal Investigator — Sinop University
Locations (2):
- Turkey (Türkiye) (2):
  - Sinop üniversitesi, Sinop
  - Sınop Univercity, Sinop

IPD SHARING:
Plan to Share IPD: No